CLINICAL TRIAL: NCT06287515
Title: Hypophysectomy by Stereotactic Radiosurgery for Cancer-Related Pain
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-0940; NCI-2024-01986 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Hypophysectomy
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- SRS hypophysectomy (Experimental): Once the radiation plan is ready, you will be brought to the radiation treatment room and positioned for treatment. You will be lying on your back on the treatment table during the radiation treatment. You will not see, hear, or feel the radiation during the treatment. The treatment time varies but may range from 1-3 three hours. Once the treatment is completed, the headframe/mask will be removed and you will be brought to a recovery area.
  Interventions: Device: Stereotactic Radiosurgery

INTERVENTIONS:
Device: Stereotactic Radiosurgery — Given by Radiation Therapy

SUMMARY:
To learn if hypophysectomy (treatment of the pituitary gland) using a type of radiation treatment called stereotactic radiosurgery (SRS) can help to relieve cancer-related pain.

DETAILED DESCRIPTION:
Primary Objective:

To determine the feasibility of enrollment and treatment of patients within MD Anderson Cancer Center with SRS hypophysectomy to plan future trials. Feasibility will be defined as completion of SRS hypophysectomy enrollment and treatment of the lead-in cohort (n=20 patients) within one year of trial activation.

Secondary Objectives:

To obtain estimates of the change from baseline over time after SRS hypophysectomy in participants with refractory cancer-related pain in the worst pain subscale of the Brief Pain Inventory (BPI) short form.57

To obtain estimates of the change from baseline over time after SRS hypophysectomy in participants with refractory cancer-related pain in the pain composite scale of the BPI short form.57

To obtain estimates of the change after SRS hypophysectomy in participants with refractory cancer-related pain in the interference scale of the BPI short form.57

To obtain estimates of the change in the daily usage of opioid medications, calculated as oral morphine equivalents (OME), over time after SRS hypophysectomy in participants with refractory cancer-related pain.

To obtain estimates of the change in mood and depressive symptoms using the Hospital Anxiety and Depression Scale (HADS) composite score over time after SRS hypophysectomy in participants with refractory cancer-related pain.60

To obtain estimates of the change in beliefs on self-efficacy using the Pain Self-Efficacy Questionnaire (PSEQ) over time after SRS hypophysectomy in participants with refractory cancer-related pain.61

To obtain estimates of the change after SRS hypophysectomy in participants with refractory cancer-related pain in quality of life as measured by the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 15 Palliative Care (QLC C15 PAL).59 To obtain estimates of neurologic toxicity related to SRS measured by the NCI's CTCAE v5.0.

Correlative Objectives:

To apply novel fMRI and DTI MRI protocols to characterize functional and connectome changes following SRS hypophysectomy.

To study neuroanatomic and histobiochemical changes of the pituitary gland/stalk after SRS hypophysectomy on post-mortem tissue.

To obtain estimates of neurocognitive changes following SRS hypophysectomy in participants with refractory cancer-related pain, including learning and memory (Hopkins Verbal Learning Test-Revised), attention (WAIS-IV Digit Span, Trail Making Test Part A, Stroop test, WAIS-IV Coding), and executive function (Trail Making Test Part B, Controlled Oral Word Association) referred to hereafter as "neurocognitive battery".63-66

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old on the day of signing informed consent and willing and able to sign a written informed consent.
* English fluency in order to complete PROs and neurocognitive assessment
* Pathologic or cytologic confirmation of malignancy.
* Poorly controlled intractable nociceptive or mixed pain limiting function or quality of life. Participants must have exhausted or not a candidate for standard of care pain control measures such as opioids, injections/ablations, conventional radiation therapy, or surgical intervention with a curative intent and pain limiting function that affects the participants quality of life in the judgment of the treating physician. Refractory status will require at least consultation and two follow-up visits with pain specialists (pain management or supportive care).
* ECOG performance status of 0-3.
* Life expectancy is greater than 4 weeks and less than 1 year in the treating physician's judgment.

Exclusion Criteria:

* Participants with prior cranial or head/neck radiation where cumulative organ-at-risk dose constraints cannot be achieved (see section 4.2).
* Inability to have an MRI of the brain for reasons such as a non-compatible bioimplant that could be displaced during MRI, shrapnel embedded (such as from war wounds), metal workers, and machinists (potential for metallic fragments in or near the eyes).
* Expressions of pain due to depression, delirium or addictive behavior
* Participants who are pregnant.
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study in the judgment of the Investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Chenyang Wang, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org